CLINICAL TRIAL: NCT00834132
Title: A Randomized, Two-Way Crossover, Single-Dose, Open-Label Study to Evaluate the Relative Bioavailability of a Test Tablet Formulation of Azithromycin (600 mg), Compared to an Equivalent Dose of a Commercially Available Reference Drug Product (Zithromax®, Pfizer, Inc.) in 24 Fed, Healthy, Adult Subjects
Brief Title: Azithromycin 600 Mg Tablets, Fed
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 02184
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Azithromycin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azithromycin (Experimental): Azithromycin 600 mg tablet (test) dosed in first period followed by Zithromax® 600 mg tablet (reference) dosed in second period
  Interventions: Drug: Azithromycin 600 mg Tablet
- Zithromax® (Active Comparator): Zithromax® 600 mg tablet (reference) dosed in first period followed by Azithromycin 600 mg tablet (test) dosed in second period
  Interventions: Drug: Zithromax® 600 mg Tablet

INTERVENTIONS:
Drug: Azithromycin 600 mg Tablet — 1 x 600mg, single-dose fed
  Arms: Azithromycin
Drug: Zithromax® 600 mg Tablet — 1 x 600mg, single-dose fed
  Arms: Zithromax®

SUMMARY:
The objective of this randomized, single-dose, two-way crossover evaluation is to compare the relative bioequivalence of a test azithromycin formulation (TEVA Pharmaceuticals USA) to an equivalent oral dose of the commercially available azithromycin (Zithromax®, Pfizer, Inc.) in a test population of 24 adult subjects under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Sex:Non-smoking Male or Female; similar proportions of each preferred.
* Age: At least 18 years.
* Weight: BMI less than 30.
* Qualifying subjects must be in good health and physical condition as determined by medical history, complete physical examination, and laboratory tests, all obtained within four (4) weeks prior to study start. The subject may not have a history of significant past illness expected to affect the investigation. The normal status of subjects will be confirmed by the following procedures:

  * Laboratory Tests: hemoglobin, hematocrit, RBC, WBC, differential count, serum electrolytes (Na, K, Cl), fasting blood glucose, BUN, bilirubin, creatinine, AST, ALT, LD, alkaline phosphatase, and urinalysis. HIV, Hepatitis B, Hepatitis C, and drugs of abuse testing will be done for screening purposes only. urine drugs of abuse testing will be repeated at each check-in. Female subjects will have a serum pregnancy test done at screening and a urine pregnancy test prior to each study period at check-in. Laboratory values which are greater than ± 20% of the normal range will not qualify unless specifically accepted (with comment) by the Principal Investigator. Results of HIV, Hepatitis B, Hepatitis C, and drugs of abuse must be negative or non-reactive for the subject to qualify for the study.
  * Electrocardiogram: A 12-lead electrocardiogram (ECG) will be obtained for all subjects. The original tracings, plus interpretation, will be included in the case report form packet.
* Subjects must read and sign the Consent Form.

Exclusion Criteria:

* Subjects not complying with the above inclusion criteria must be excluded from the study.
* In addition, any one of the conditions listed below will exclude a subject from the study:

  * History of treatment for alcoholism, substance abuse, or drug abuse within past 24 months.
  * History of malignancy, stroke, diabetes, cardiac, renal or liver disease, or other serious illness.
  * History of treatment for asthma within the past five (5) years.
  * History of treatment for any gastrointestinal disorder within the past five (5) years.
  * History of hepatic function impairment.
  * Females who are pregnant or lactating.
  * History of hypersensitivity to azithromycin, erythromycin, or any macrolide antibacterial agent.
* Conditions upon screening which might contraindicate or require that caution be used in the administration of azithromycin, including:

  * Sitting systolic blood pressure below 90 mmHg, or diastolic pressure below 50 mmHg.
  * Heart rate less than 50 beats per minute after a 5-minute rest in a seated position.
* Inability to read and/or sign the consent form.
* Treatment with any other investigational drug during the four (4) weeks prior to the initial dosing for this study.
* Subjects who have donated blood within four (4) weeks prior to the initial dosing for this study.
* Subjects who smoke or use tobacco products or are currently using nicotine products (patches, gums, etc.) At least three (4) consecutive months of abstinence is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-07; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Azber Ansar, M.D., Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Gateway Medical Research, Inc., Saint Charles, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin (Test) First: Azithromycin 600 mg tablet (test) dosed in first period followed by Zithromax® 600 mg tablet (reference) dosed in second period
- Zithromax® (Reference) First: Zithromax® 600 mg tablet (reference) dosed in first period followed by Azithromycin 600 mg tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Azithromycin (Test) First | Zithromax® (Reference) First
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout: 21 Days
Arm/Group | Azithromycin (Test) First | Zithromax® (Reference) First
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Azithromycin (Test) First | Zithromax® (Reference) First
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin (Test) First | Zithromax® (Reference) First | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 8 | 7 | 15
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 7 | 9 | 16
  Black | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration - Azithromycin in Plasma
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 168 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Azithromycin: Azithromycin 600 mg tablet (test) dosed in either period
- Zithromax®: Zithromax® 600 mg tablet (reference) dosed in either period
Arm/Group | Azithromycin | Zithromax®
Number analyzed (Participants) | 24 | 24
ng/mL | 561.556 (199.349) | 592.311 (255.261)
Statistical Analysis 1: Comparison: Azithromycin vs Zithromax®; Test type: Non-Inferiority or Equivalence — Using PROC GLM procedures in SAS, analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Test/Ref Ratio of LS Means x 100 = 94.81, 90% CI [84.77 to 106.04] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated) - Azithromycin in Plasma
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 168 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Azithromycin | Zithromax®
Number analyzed (Participants) | 24 | 24
ng*h/mL | 7025.920 (1583.546) | 6964.092 (1621.163)
Statistical Analysis 1: Comparison: Azithromycin vs Zithromax®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 100.89, 90% CI [96.00 to 106.03] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)- Azithromycin in Plasma
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 168 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Azithromycin | Zithromax®
Number analyzed (Participants) | 24 | 24
ng*h/mL | 6132.710 (1483.937) | 6063.795 (1436.447)
Statistical Analysis 1: Comparison: Azithromycin vs Zithromax®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 101.14, 90% CI [96.05 to 106.49] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.